CLINICAL TRIAL: NCT04423029
Title: A Phase 1/1b, First-In-Human, Multi-Part, Open-Label, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of DF6002 as a Monotherapy and in Combination With Nivolumab in Patients With Locally Advanced or Metastatic Solid Tumors, and Expansion in Selected Indications
Brief Title: A Study of DF6002 Alone and in Combination With Nivolumab
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dragonfly Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF6002 - 001; 2023-510511-19 (EudraCT Number)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors
Keywords: Advanced or Metastatic Solid Tumors; Melanoma; Non-small Cell Lung Cancer; Nivolumab; DF6002
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation / Monotherapy / Subcutaneously or Intravenously (Experimental): Subcutaneous portion of the study is complete. Dosing DF6002 Q4W
  Interventions: Drug: DF6002
- Dose Escalation / Combination / Subcutaneously or Intravenously (Experimental): Subcutaneous portion of the study is complete. Dosing DF6002 Q4W Dosing nivolumab Q4W
  Interventions: Drug: DF6002; Drug: Nivolumab
- Safety/PK/PD / Monotherapy / Subcutaneously or Intravenously (Experimental): Subcutaneous portion of the study is complete. Dosing DF6002 Q4W
  Interventions: Drug: DF6002
- Safety/PK/PD / Combination / Subcutaneously or Intravenously (Experimental): Subcutaneous portion of the study is complete. Dosing DF6002 Q4W Dosing nivolumab Q4W
  Interventions: Drug: DF6002; Drug: Nivolumab
- Efficacy Expansion / Combination / Subcutaneously or Intravenously / Melanoma (Experimental): Subcutaneous portion of the study is complete. 2L+ melanoma Dosing DF6002 Q4W Dosing nivolumab Q4W
  Interventions: Drug: DF6002; Drug: Nivolumab
- Efficacy Expansion / Combination / Subcutaneously or Intravenously / Non-Melanoma (Experimental): Subcutaneous portion of the study is complete. 2L+ non-melanoma skin cancer (including cSCC, BCC, and MCC) Dosing DF6002 Q4W Dosing nivolumab Q4W
  Interventions: Drug: DF6002; Drug: Nivolumab

INTERVENTIONS:
Drug: DF6002 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Dose Escalation / Combination / Subcutaneously or Intravenously; Efficacy Expansion / Combination / Subcutaneously or Intravenously / Melanoma; Efficacy Expansion / Combination / Subcutaneously or Intravenously / Non-Melanoma; Safety/PK/PD / Combination / Subcutaneously or Intravenously

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug-levels, drug-effects and preliminary anti-tumor activity of DF6002 alone and in combination with Nivolumab in participants with advanced solid tumors.

DETAILED DESCRIPTION:
Assess the safety and tolerability of subcutaneous (SC) and intravenous (IV) administration of DF6002, as monotherapy and in combination with nivolumab, and to determine the maximum tolerated dose (MTD) and recommended efficacy expansion dose (REED) of SC and IV DF6002, both as monotherapy and in combination with nivolumab, for patients with advanced (unresectable, recurrent, or metastatic) solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic solid tumors, for which no standard therapy exists or standard therapy has failed among the following tumor types: melanoma, non-small cell lung cancer, small cell lung cancer, head and neck squamous cell, urothelial, gastric, esophageal, cervical, hepatocellular, merkel cell, cutaneous squamous cell carcinoma, renal cell, endometrial, triple-negative breast, ovarian, and prostate
* ECOG performance status of 0 or 1
* Clinical or radiological evidence of disease
* Adequate hematological, hepatic and renal function
* Anticoagulants are required for the following: Khorana Risk Score ≥ 2 or as assessed by Investigator as being at high risk for venous thromboembolism (VTE) or history of VTE ≥ 6 months from enrollment

Exclusion Criteria:

* Concurrent anticancer treatment (with the exception of palliative bone directed radiotherapy), immune therapy, or cytokine therapy (except for erythropoietin), major surgery (excluding prior diagnostic biopsy), concurrent systemic therapy with steroids or other immunosuppressive agents, or use of any investigational drug within 28 days before the start of study treatment
* Prior treatment with DF6002, recombinant human interleukin-12 (rhIL-12)-directed therapy, or any drug containing an interleukin-12 (IL-12) moiety
* Previous malignant disease other than the current target malignancy within the last 3 years, with the exception of basal or squamous cell carcinoma of the skin, localized prostate cancer or cervical carcinoma in situ
* Rapidly progressive disease
* Serious cardiac illness or medical conditions
* Known diagnosis of antiphospholipid syndrome or clinically significant hereditary thrombophilia

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | During the first 3 weeks of treatment
  Dose Escalation
Overall Response Rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per an Independent Endpoint Review Committee (IERC) | Up to 2 years
  Efficacy Expansion Arms

SECONDARY OUTCOMES:
Amount of Treatment Emergent Adverse Events (TEAEs) | Up to 2 years
  Number of participants with TEAEs
Severity of TEAEs | Up to 2 years
  Severity of the TEAEs seen in study participants
Duration of TEAEs | Up to 2 years
  How long the TEAEs seen last
Number of participants with changes from baseline in clinical laboratory parameters | Up to 2 years
  Overall change, if any, after treatment
Number of participants with changes from baseline in electrocardiogram (ECG) parameters | Up to 2 years
  Overall change, if any, after treatment
Number of participants with changes from baseline in vital sign parameters | Up to 2 years
  Overall change, if any, after treatment
Duration of Response (DOR) according to RECIST 1.1 per Investigator assessment | Up to month 24
  Overall change, if any, after treatment
Area under the plasma concentration-time curve from the time of dosing to the time of the last observation (AUC 0-T) | Up to day 28
  Overall change, if any, after treatment
Area under the plasma concentration-time curve from the time of dosing extrapolated to infinity (AUC 0-INF) | Up to day 28
  Overall change, if any, after treatment
Maximum serum concentration observed post-dose (Cmax) | Up to day 28
  Overall change, if any, after treatment
Best overall response (BOR) according to RECIST 1.1 per Investigator assessment | Approximately one year
  Overall change, if any, after treatment
Clinical benefit rate (CBR) according to RECIST 1.1 per Investigator assessment | Up to 2 years
  Overall change, if any, after treatment
Confirmed ORR per RECIST 1.1 per Investigator assessment | Up to 2 years
  Phase 1/1b only
Progression-free survival (PFS) according to RECIST 1.1 per Investigator assessment | Up to 2 years
  Phase 2 only
CBR according to RECIST 1.1 per IERC | Up to 2 years
  Phase 2 only
PFS according to RECIST 1.1 per IERC | Up to 2 years
  Phase 2 only
DOR according to RECIST 1.1 per IERC | Up to month 24
  Phase 2 only
Unconfirmed response after 4 cycles according to RECIST 1.1 | Up to 2 years
  Phase 2 only
Overall Survival (OS) | Up to 5 years
  Phase 2 only
Serum titers of anti-DF6002 antibodies | Up to 2 years
  Phase 2 only
Serum titers of anti-nivolumab antibodies | Up to 2 years
  Phase 2 only

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Dragonfly Therapeutics
Locations (32):
- United States (21):
  - University of California Irvine, Orange, California
  - SCRI - HealthOne Denver, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Local Institution, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - SCRI - Tennessee Oncology - Saint Thomas West Clinic, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute and Hospital, Salt Lake City, Utah
  - USOR - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (2):
  - Local Institution - 0023, Box Hill
  - Local Institution - 0022, Heidelberg
- France (4):
  - Institut Bergonié, Bordeaux
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - START Madrid - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona